CLINICAL TRIAL: NCT05290883
Title: Antithrombotic Activities of a Novel Yoghurt Drink: a Postprandial Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Principal Investigator, Ioannis Zabetakis, Senior Lecturer, University of Limerick
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S&E REC No. 2022_01_01_S&E
Record Dates: First submitted 2022-03-04; First posted 2022-03-22 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group A: Yoghurt drink (polar lipid) intervention (Experimental)
  Interventions: Dietary Supplement: Novel yoghurt drink containing Polar Lipids

INTERVENTIONS:
Dietary Supplement: Novel yoghurt drink containing Polar Lipids — Postprandial decreased platelet activation/aggregation in subjects, after the yoghurt drink consumption

SUMMARY:
The project aims to investigate the antithrombotic activity of the novel yoghurt drink enriched with polar lipids derived from ovine milk. The health claims the formulated novel or functional food on EFSA guidelines "The scientific requirements for health claims related to antioxidants, oxidative damage and cardiovascular health" and in a particular paragraph 5.4, "Claims on reduced platelet aggregation" "Platelet hyperactivity and hypercoagulability states are more commonly observed in subjects with cardiovascular (CV) risk factors. Healthy subjects or participants at very low risk of CV disease normally have non-activated circulating platelets. Reducing platelet aggregation in subjects with platelet activation during sustained exposure to the food/constituent (e.g., four weeks) would be a beneficial physiological effect".

Within this investigation, the postprandial effects of this novel yoghurt drink against platelet aggregation are going to be studied ex vivo in blood from healthy human subjects as described in previously established procedures.

ELIGIBILITY:
Inclusion Criteria:

* • Healthy subjects need to have their dietary and dairy intake within the range [1-2 serves per week]

Exclusion Criteria:

* Subjects will be excluded from the study if they are

  * Under medication and intake of dietary supplements
  * Treatment for blood clotting disorders or dyslipidaemia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2021-07-18 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
An investigation of anti-platelet or antithrombotic effect of novel yoghurt drink by platelet aggregometry | 0 mins (preprandially) to 240 mins (postprandially)
  An investigation of anti-platelet or antithrombotic effect of novel yoghurt drink by platelet aggregometry will be carried out. The postprandial effect of novel yoghurt drink will be studied by using a platelet aggregation method as per literature. The antithrombotic effect of yoghurt drink lipids will be studied, using PAF and TRAP as platelet aggregation mediators. The investigation will be based on the study-specific platelet aggregometry analysis. Subjects will come to the lab after overnight fasting and they will be provided yoghurt drink (200mL); the activation of their platelets will be monitored over a period of 4 hours (0 to 4 hours study with 1 hour check points).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsoupras A, Zabetakis I, Lordan R. Platelet aggregometry assay for evaluating the effects of platelet agonists and antiplatelet compounds on platelet function in vitro. MethodsX. 2018 Dec 26;6:63-70. doi: 10.1016/j.mex.2018.12.012. eCollection 2019. PMID 30619728
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30619728/